CLINICAL TRIAL: NCT04714827
Title: A Clinical Study to Evaluate the Safety and Effectiveness of CD19-BCMA CAR-T Cells Immunotherapy in Patients With Relapsed or Refractory Multiple Myeloma
Brief Title: Targeting CD19 and BCMA CAR-T Cells Immunotherapy in Patients With Relapsed or Refractory Multiple Myeloma
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanxi Province Cancer Hospital (Other)
Collaborators: Novatim Immune Therapeutics (Zhejiang) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CAR-T SXZL03
Record Dates: First submitted 2021-01-07; First posted 2021-01-19 (Actual); Last update posted 2023-12-29 (Actual); Status verified 2023-12

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Low Dose Group (Experimental): KQ-2003 CAR-T cells injection, infused only once,3-6 subjects of low dose group will be intravenously infuse with 1.0×10^6 CAR+T cells/kg.
  Interventions: Biological: KQ-2003 CAR-T cells
- Middle Dose Group (Experimental): KQ-2003 CAR-T cells injection, infused only once,3-6 subjects of low dose group will be intravenously infuse with 2.5×10^6 CAR+T cells/kg.
  Interventions: Biological: KQ-2003 CAR-T cells
- High Dose Group (Experimental): KQ-2003 CAR-T cells injection, infused only once,3-6 subjects of low dose group will be intravenously infuse with 5.0×10^6 CAR+T cells/kg.
  Interventions: Biological: KQ-2003 CAR-T cells
- Amplification Dose Group (Experimental): KQ-2003 CAR-T cells injection, infused only once.After determined maximum tolerated dose,15 subjects of amplification dose group will be intravenously infuse with 1.0-5.0×10^6 CAR+Tcells/kg.
  Interventions: Biological: KQ-2003 CAR-T cells

INTERVENTIONS:
Biological: KQ-2003 CAR-T cells — A autologous doping CAR - T cells injection targets with CD19 and BCMA，fluorine dara marina injection(30 mg/m2，QD×3d) and cyclophosphamide injection (300 mg/m2，QD×3d)will be used to remove the lymphocyte before infusion KQ-2003 CAR-T cells .
  Other Names: Fluorine dara marina injection; Cyclophosphamide injection; CD19-BCMA CAR-T Cells

SUMMARY:
Evaluation the safety,tolerability, preliminary efficacy,and PK/PD of KQ-2003 CAR-T cells for the treatment of multiple myeloma

DETAILED DESCRIPTION:
A non randomized study ,plans to enrollment 24 patients of B cell lymphoma ，divided into low, medium and high dose groups，to evaluate the safety and tolerability of KQ-2003 CAR-T cells immunotherapy in patients with relapsed or refractory B cell lymphoma ，to evaluate the preliminary efficacy and observe PK/PD parameters of KQ-2003 CAR-T cells immunotherapy in patients with relapsed or refractory multiple myeloma .

ELIGIBILITY:
Inclusion Criteria:

1. Agreed to participate in this study and signed informed consent, and willing to finish all the test procedure.
2. Age ≧ 18 years of age, gender not limited;
3. According to IMWG， diagnosis of multiple myeloma patients;
4. ECOG physical score ≤2 points ;
5. Relapsed multiple myeloma: disease progressed after received at least 3 lines treatment (must including the proteasome inhibitors and immune modulators); Refractory multiple myeloma: early treatment has never reached more than MR and curative effect; Or early treatment has reached more than MR and curative effect, but the subsequent treatment process or disease progress within 60 days after the last treatment ;
6. Have a measurable lesions in screening period (conform to one of the following standards: (1) the serum M protein: IgG protein≥10g/L, or IgA M protein ≥5g/L, or IgD M protein ≥5g/L; (2) M protein urine ≥200mg/24h; (3)If M protein in serum or urine cannot be measured,under the condition of the abnormal serum free light chain ratio,serum free light chain immunoglobulin or 100 mg/L;
7. Test results in screening period: (1) Hb≥60 g/L (7 days before the inspection without blood transfusion),PLT≥ 50 x 10 ^ 9 / L(7 days before the inspection without blood transfusion) ,ALC≥0.3×10^9/L,ANC≥0.75×10^9/L; (2)AST≤3ULN,ALT≤3ULN,TBIL≤2ULN；Ccr≥30 mL/min/1.73 m2;Correction of serum calcium ≤3.1mmol/L（≤12.5mg/dL）; LVEF≥40%； Baseline peripheral blood oxygen saturation ≥95%;
8. Female subjects with fertility ,pregnancy blood test results should be negative in screening period and before remove the lymphocyte ;
9. Expected to survival more than 3 months;

Exclusion Criteria:

1. The active hepatitis b, HBV - DNA detection lower limit of the subjects above research center; Hepatitis c virus (HCV) antibody positive and peripheral blood HCV - RNA positive subjects; Antibodies to HIV positive subjects; Early syphilis screening antibody positive;
2. The other clinical significance of active virus, bacterial infection, or failing to control systemic fungal infection;
3. Any instability of systemic disease, including but not limited to, unstable angina, cerebrovascular accident, or transient ischemic (within 6 months prior to screening), myocardial infarction (within 6 months prior to screening), New York heart association (NYHA) classification level III or higher congestive heart failure, drug control of serious arrhythmia, liver, kidney or metabolic diseases, as well as the standard treatment cannot control high blood pressure;
4. In past two years, because of autoimmune diseases such as crohn's disease, rheumatoid arthritis and systemic lupus erythematosus (sle), etc.) causing end-organ damage, or need systemic application of immunosuppressive drugs;
5. Had a history of the central nervous system diseases, such as epilepsy, serious brain damage, dementia, Parkinson's disease, psychosis,etc which influence the appraising of test,;
6. Diagnosed with other active malignancy in past five years(the basal or scaly skin cancer, superficial bladder cancer, breast cancer in situ, which has been cured and does not require follow-up treatment are not included );
7. Known allergic to cyclophosphamide, fluorine dara marina or CAR - T cell s including accessories, DMSO ;
8. Patients with pregnancy or lactation, patients do not want to take effective contraceptive measures within 6months after infusion CAR-T cells;
9. The other situations that researchers determined doesn't fit to participate in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2021-01-22 (Actual); Primary Completion 2024-09-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
DLT | Form infusion CAR-T cells to 28 days after infusion
  Observe wether dose limiting toxicity will happened in dose escalation phase
ORR | Form infusion CAR-T cells to 2 years after infusion
  The overall response rate after CAR-T Cells immunotherapy

SECONDARY OUTCOMES:
Incidence of various types of adverse recation | Form infusion CAR-T cells to 2 years after infusion
  According to CTCAE 5.0, record the level , type of adverse events, evaluat the correlation of CD19-BCMA CAR-T cells
PFS | Form infusion CAR-T cells to 2 years after infusion
  Progression-free surial
DOR | Form infusion CAR-T cells to 2 years after infusion
  Duration of Response
OS | Form infusion CAR-T cells to subjects died，assessed up to 60 months
  Overall survival
Cmax | Before removal of lymphocytes, before CAR - T cells infusion, Day1, Day3, Day5, Day7, Day10, Day14, Day21, Day28, Month2, Month3, Month6, Month9, Month12, Month15, Month18, Month21, Month24
  By measuring the CAR - T cells copy number and the positive rate, peak plasma concentration is determined
Tmax | Before removal of lymphocytes, before CAR - T cells infusion, Day1, Day3, Day5, Day7, Day10, Day14, Day21, Day28, Month2, Month3, Month6, Month9, Month12, Month15, Month18, Month21, Month24
  The maximum concentration of time
AUC（0-720d） | Before removal of lymphocytes, before CAR - T cells infusion, Day1, Day3, Day5, Day7, Day10, Day14, Day21, Day28, Month2, Month3, Month6, Month9, Month12, Month15, Month18, Month21, Month24
  Area under the plasma concentration versus time curve
Concentration of IL2 level | Before removal of lymphocytes, before CAR - T cells infusion, Day1, Day3, Day5, Day7, Day10, Day14, Day21, Day28, Month2, Month3, Month6, Month9, Month12, Month15, Month18, Month21, Month24
  The levels of cytokines（IL2 ）in peripheral blood and bone marrow
Concentration of IL6 level | Before removal of lymphocytes, before CAR - T cells infusion, Day1, Day3, Day5, Day7, Day10, Day14, Day21, Day28, Month2, Month3, Month6, Month9, Month12, Month15, Month18, Month21, Month24
  The levels of cytokines（ IL6 ）in peripheral blood and bone marrow
Concentration of IL10 level | Before removal of lymphocytes, before CAR - T cells infusion, Day1, Day3, Day5, Day7, Day10, Day14, Day21, Day28, Month2, Month3, Month6, Month9, Month12, Month15, Month18, Month21, Month24
  The levels of cytokines（IL10 ）in peripheral blood and bone marrow
Concentration of TNF-α level | Before removal of lymphocytes, before CAR - T cells infusion, Day1, Day3, Day5, Day7, Day10, Day14, Day21, Day28, Month2, Month3, Month6, Month9, Month12, Month15, Month18, Month21, Month24
  The levels of cytokines（TNF-α ）in peripheral blood and bone marrow
Concentration of IFN-γ level | Before removal of lymphocytes, before CAR - T cells infusion, Day1, Day3, Day5, Day7, Day10, Day14, Day21, Day28, Month2, Month3, Month6, Month9, Month12, Month15, Month18, Month21, Month24
  The levels of cytokines（IFN-γ ）in peripheral blood and bone marrow

CONTACTS AND LOCATIONS:
Overall Officials: Liping Su, M.D., Principal Investigator — Hematology Department of ShanXi Cancer Hospital
Locations (1):
- Hematology Department of ShanXi Cancer Hospital, Taiyuan, Shanxi, China

IPD SHARING:
Plan to Share IPD: Yes
Plan to Share Clinical Study Report within six months after the study completed
Supporting Information: CSR
Time Frame: Within six months after the study completed
Access Criteria: Research site